CLINICAL TRIAL: NCT03628482
Title: A Randomized Controlled Study to Compare Efficacy of Continuous Versus Pulsed Radiofrequency Treatment of Genicular Nerves to Alleviate Pain and Improve Functional Impairment in Patients With Advanced Osteoarthritis of the Knee
Brief Title: Pulsed Radiofrequency to Relieve Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gasthuis Zusters Antwerpen (Other)
Collaborators: ZOL (Other); Hospital General de Jerez de la Frontera (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MMSP-LV2
Record Dates: First submitted 2018-08-06; First posted 2018-08-14 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Pain Syndrome
MeSH Terms: conditions — Somatoform Disorders | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned using a computer-generated randomization schedule to receive percutaneous radiofrequency treatment of the genicular nerves that was administered in either the continuous or in the pulsed mode.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were randomly assigned using a computer-generated randomization schedule to receive either continuous or pulsed radiofrequency treatment of genicular nerves. The allocation sequence was concealed from the researcher enrolling and assessing participants in sequentially numbered, opaque, sealed and stapled envelopes. The corresponding envelopes were opened only at the time of intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CRF group (Active Comparator): Patients were assigned to receive continuous radiofrequency (CRF) treatment of genicular nerves
  Interventions: Procedure: CRF
- PRF group (Experimental): Patients were assigned to receive pulsed radiofrequency (CRF) treatment of genicular nerves
  Interventions: Procedure: PRF

INTERVENTIONS:
Procedure: CRF — For continuous radiofrequency ablation the electrode tip temperature was raised to 80°C during 90 s.
  Other Names: Continuous radiofrequency treatment
  Arms: CRF group
Procedure: PRF — The procedure for PRF is almost identical to that applied for CRF, except that the current is typically carried out in 20 ms pulses every 0.5 s at a temperature that does not exceed 42 °C during 360 s.
  Other Names: Pulsed radiofrequency treatment
  Arms: PRF group

SUMMARY:
Knee osteoarthritis is a leading cause of chronic pain, disability, and decreased quality of life. Lesioning of genicular nerves by continuous radiofrequency treatment proved to be effective in relieving pain and disability caused by osteoarthritis of the knee. In contrast to continuous radiofrequency lesioning, pulsed radiofrequency treatment offers pain control with no or only minimal histological lesions. As a non-destructive alternative to continuous radiofrequency ablation, pulsed radiofrequency treatment may have inherent appeal because it may mitigate concerns regarding complications associated with the ablation of nerves. However, studies comparing the ability of the continuous and the pulsed modalities of radiofrequency treatment to relieve pain and incapacity due to osteoarthritis of the knee are lacking. Therefore, it was the aim of the investigators of current study to compare efficacy of continuous and pulsed radiofrequency treatments of genicular nerves to alleviate pain and disability in patients with advanced osteoarthritis of the knee.

DETAILED DESCRIPTION:
Following approval of the Regional Research Ethics Committee written informed consent was obtained from all patients. Current randomized controlled trial included patients with grade 3-4 gonarthritis suffering from intractable knee pain, scoring ≥5 on the Visual Analog Scale (VAS) during >6 months. Therapy was based on ultrasound guided radiofrequency treatment of the superior medial, superior lateral and inferior medial genicular nerves. VAS and Western Ontario and MacMaster Universities Osteoarthrosis (WOMAC) scores were assessed before therapy and at 1, 6 and 12 months following intervention. Eligible patients were randomized in two treatment groups according to the modality of radiofrequency current to which targeted genicular nerves had to be exposed, i.e, the pulsed and the continuous radiofrequency groups. Both two way repeated measures analysis of variance and generalized estimating equations were used to determine whether the VAS and WOMAC scores obtained with either the continuous or the pulsed radiofrequency modalities at each of the 4 times of assessment, i.e. at pre-treatment control and at 1, 6 and 12 months after the intervention, were different.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients suffered from chronic pain (during>6months) of moderate to severe intensity (scoring ≥5 on a 0- to 10-point continuous visual analog scale [VAS] ranging from none [0] to an extreme amount of pain [10]) due to advanced osteoarthritis of the knee (grades 3-4 according to the Kellgren-Lawrence classification. The pain proved to be resistant to conservative treatments including physiotherapy, oral analgesics, and intraarticular injection with hyaluronic acids or steroids. In this study, genicular nerve ablation was applied as an alternative analgesic approach for those who refused knee arthroplasty; were judged by their surgeons as being inappropriate for surgical treatment, for example, because of cardiovascular or other comorbidities; or who had to be managed for persistent pain and stiffness after total knee arthroplasty.

Exclusion Criteria:

* The exclusion criteria included knee-pain related disorders that might benefit from other interventions, for example, patellofemoral disorders, meniscal injuries, ligamentous laxity, and so on, acute knee pain associated with radicular neuropathy or intermittent claudication, connective tissue diseases, serious neurologic or psychiatric disorders, mental deterioration impeding adequate communication or collaboration, anticoagulant medications, pacemakers, prior electroacupuncture treatment, and injection with steroids or hyaluronic acids during the previous 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) score | VAS score at 12 months following the radiofrequency treatment.
  The pain VAS is a unidimensional measure of pain intensity (1), rated on a continuous scale which is 10 centimeters in length, and anchored by 2 verbal descriptors, one for each symptom extreme , " no pain " and " worst imaginable pain ". Our null hypothesis was that no significant difference would exist in VAS scores between the continuous and the pulsed radiofrequency groups at 12 months following the intervention.

SECONDARY OUTCOMES:
The Western Ontario and Mac Master Universities Osteoarthritis Index (WOMAC) | WOMAC score at 12 months following the radiofrequency treatment.
  The Western Ontario and Mac Master Universities Osteoarthritis Index (WOMAC) is a standardized questionnaire used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. Our null hypothesis was that no significant difference would exist in the WOMAC scores between the continuous and the pulsed radiofrequency groups at 12 months following the intervention.
Adverse events | adverse effects at 12 months following the radiofrequency treatment.
  Adverse effects including abnormal proprioception, numbness, paresthesia, neuralgia, and motor weakness were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Zundert, Principal Investigator — ZOL
Locations (1):
- Luc Vanlinthout, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
IPD will be shared when current study has been published

REFERENCES:
- [Derived] Santana-Pineda MM, Vanlinthout LE, Santana-Ramirez S, Vanneste T, Van Zundert J, Novalbos-Ruiz JP. A Randomized Controlled Trial to Compare Analgesia and Functional Improvement After Continuous Neuroablative and Pulsed Neuromodulative Radiofrequency Treatment of the Genicular Nerves in Patients with Knee Osteoarthritis up to One Year After the Intervention. Pain Med. 2021 Mar 18;22(3):637-652. doi: 10.1093/pm/pnaa309. PMID 33179073